CLINICAL TRIAL: NCT01743404
Title: Double-blinded Placebo-controlled Multicenter Study of Anti-atherosclerotic Activity of Inflaminat in Asymptomatic Participants With Subclinical Atherosclerosis
Brief Title: Study of Anti-atherosclerotic Activity of Inflaminat in Asymptomatic Participants With Subclinical Atherosclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Atherosclerosis Research, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IAR-INFL
Record Dates: First submitted 2012-12-02; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-09

CONDITIONS: Carotid Atherosclerosis
Keywords: atherosclerosis; inflammation; intima-media thickness
MeSH Terms: conditions — Carotid Artery Diseases; Atherosclerosis; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inflaminat (Active Comparator): Inflaminat 500 mg tablet by mouth three times a day
  Interventions: Dietary Supplement: Inflaminat
- Sugar pill (Placebo Comparator): Placebo 500 mg tablet by mouth three times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Inflaminat
  Arms: Inflaminat
Drug: Placebo — Sugar pill manufactured to mimic Inflaminat 500 mg tablet
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to investigate the anti-atherosclerotic effect of long-term anti-inflammatory therapy (Inflaminat) in asymptomatic participants with subclinical atherosclerosis of carotid arteries.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 40 to 70 years
* Subclinical carotid atherosclerosis detected by B-mode ultrasound (increased intima-media thickness 1000-2000 mcm)
* Arterial normotension or mild arterial hypertension (systolic blood pressure <160 mm Hg, diastolic blood pressure <90 mm Hg)
* Absence of chronic diseases demanding permanent drug administration (more than 2 month per year)

Exclusion Criteria:

* Personal history of stroke or transient ischemic attacks
* Chronic diseases demanding drug administration more than during 2 month per year
* Individual intolerance of Inflaminat or appearance of side effects

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-09; Primary Completion 2013-02 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
B-mode ultrasound of carotid arteries | up to 2 years
  Variation of intima-media thickness of common carotid arteries

SECONDARY OUTCOMES:
Measure of serum atherogenicity | up to 2 years
  Change of the ability of serum to induce cholesterol accumulation in cultured cells

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Atherosclerosis Research, Moscow, Moscow, Russia